CLINICAL TRIAL: NCT04277845
Title: Randomized Phase II Study of Bortezomib, Lenalidomide and Dexamethasone Versus Lenalidomide and Dexamethasone in Elderly Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Randomized Phase II Study in Elderly Patients With Newly Diagnosed Multiple Myeloma
Acronym: KMM1910
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kihyun Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2019-08-025
Record Dates: First submitted 2020-02-16; First posted 2020-02-20 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1: 1 cycle will be repeated every 4 weeks
  Bortezomib 1.3mg/m2 SC D1, 8, 15 - Dose adjustment for more than 85 : 1.0mg/m2 SC D1, 8, 15
  Lenalidomide 25mg/d D1-21
  - Dose adjustment for more than 75 : 15mg/d D1-21
  Dexamethasone 40mg D1, 8, 15, 22 - Dose adjustment for more than 75 years old: 20mg If it is difficult to maintain bortezomib due to unacceptable toxicity, it can early discontinue from Group 1.
  <for patients with old age or frail>
  Bortezomib 1.0mg/m2 SC D1, 8, 15
  : Dose adjustment for more than 85 : 1.0mg/m2 SC D1,8,15 Lenalidomide 15mg/d D1-21 Dexamethasone 20mg D1, 8, 15, 22
  Interventions: Drug: Bortezomib, Lenalidomide, Dexamethasone
- Group 2 (Active Comparator): Group 2: 1 cycle will be repeated every 4 weeks
  Lenalidomide 25mg/d D1-21
  * Dose adjustment for more than 75: 15mg Dexamethasone 40mg D1, 8, 15, 22
  * Dose adjustment for more than 75: 20mg
  <for patients with old age or frail>
  1. Lenalidomide 15mg/d D1-21
  2. Dexamethasone 20mg D1, 8, 15, 22
  Interventions: Drug: Bortezomib, Lenalidomide, Dexamethasone

INTERVENTIONS:
Drug: Bortezomib, Lenalidomide, Dexamethasone — Bortezomib, Lenalidomide and Dexamethasone versus Lenalidomide and Dexamethasone
  Other Names: Lenalidomide, Dexamethasone

SUMMARY:
To compare the efficacy and safety of bortezomib, lenalidomide and dexamethasone in elderly frail patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
Group 1: 1 cycle will be repeated every 4 weeks

1. Bortezomib 1.3mg/m2 SC D1, 8, 15

   - Dose adjustment for more than 85 : 1.0mg/m2 SC D1, 8, 15
2. Lenalidomide 25mg/d D1-21

   - Dose adjustment for more than 75 : 15mg/d D1-21
3. Dexamethasone 40mg D1, 8, 15, 22

   * Dose adjustment for more than 75 years old: 20mg
   * If it is difficult to maintain bortezomib due to unacceptable toxicity, it can early discontinue from Group 1.

<for patients with old age or frail>

1. Bortezomib 1.0mg/m2 SC D1, 8, 15 : Dose adjustment for more than 85 : 1.0mg/m2 SC D1,8,15
2. Lenalidomide 15mg/d D1-21
3. Dexamethasone 20mg D1, 8, 15, 22

Group 2: 1 cycle will be repeated every 4 weeks

1. Lenalidomide 25mg/d D1-21 - Dose adjustment for more than 75: 15mg
2. Dexamethasone 40mg D1, 8, 15, 22 - Dose adjustment for more than 75: 20mg <for patients with old age or frail>

1) Lenalidomide 15mg/d D1-21 2) Dexamethasone 20mg D1, 8, 15, 22

ELIGIBILITY:
[Inclusion criteria]

1. Newly diagnosed with multiple myeloma
2. Older than 70 years
3. Ineligible for autologous stem cell transplantation
4. No history of prior treatment for multiple myeloma
5. At least one of the following measuarble disease

   * Serum M-protein ≥ 0.5 g/dL, or urine M-protein ≥ 200mg/24 hour, or
   * In patients without detectable serum or urine M-protein, serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal serum kappa/lambda ratio.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
7. Adequate hepatic functionwith bilirubin < 1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the ULN.
8. Left ventricular ejection fraction (LVEF) ≥ 40%.
9. *Absolute Neutrophil Count (ANC) ≥ 1000/mm³: Screening ANC should be independent of growth factor support for ≥ 1 week;

   * Hemoglobin ≥ 8.0 g/dL (Use of erythropoietic stimulating factors and red blood cell transfusions is allowed);
   * Platelet count ≥ 50,000/mm³ (≥ 30,000/mm³ -if myeloma involvement in the bone marrow is >50%): Patients should not have received platelet transfusions
   * for at least 1 week prior to obtaining the screening platelet count.
10. Calculated or measured creatinine clearance (CrCl) of ≥ 15 mL/min

    - Calculation should be based on standard formula such as the Cockcroft and Gault: [(140 - Age) x Mass (kg) / (72 x Creatinine mg/dL)]; multiply result by 0.85 if female.
11. Written informed consent in accordance with institutional guidelines.
12. Female patients of child-bearing potential (FCBP) must have two negative pregnancy tests (sensitivity of at least 25 mIU/mL) prior to starting lenalidomide. The first pregnancy test must be performed within 10 to 14 days prior to the start of lenalidomide and the second pregnancy test must be performed within 24 hours prior to the start of lenalidomide.

    Effective method of contraception should be used during and for 28 days following last dose of drug

    - FCBP is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
13. Male patients must use an effective barrier method of contraception during study and for 28 days following the last dose if sexually active with a FCBP.

[Exclusion criteria]

1. Relapsed or refractory multiple myeloma
2. Multiple Myeloma of IgM subtype.
3. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
4. Plasma cell leukemia or circulating plasma cells ≥ 2 × 10^9/L.
5. Waldenstrom's Macroglobulinemia.
6. Patients with known amyloidosis.
7. Patients got approved chemotherapy or investigational anticancer therapeutics within 21 days prior to the 1st day of 1st cycle.
8. Focal radiation therapy within 7 days prior to the 1st day of 1st cycle.
9. Immunotherapy within 21 days prior to the 1st day of 1st cycle.
10. Major surgery (excluding kyphoplasty) within 28 days prior to 1st day of 1st cycle.
11. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within four months prior to 1st day of 1st cycle.
12. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents within 14 days prior to 1st day of 1st cycle.
13. Known human immunodeficiency (HIV) seropositive, hepatitis C infection, and/or hepatitis B (But, allow the patient who is DNA(-) or responding to antiviral therapy even if patient is HBsAg(+) or anti-HBc(+)).
14. Patients with known cirrhosis.
15. Female patients who are pregnant or lactating.
16. Patients with contraindication to dexamethasone.
17. Hypersensitivity to antiviral drugs, Contraindication to any of the required concomitant drugs or supportive treatments due to preexisting pulmonary or cardiac impairment.
18. Patients with end-stage renal disease requiring hemodialysis or peritoneal dialysis
19. Patients with a history of malignant tumors other than the target disease, except for the following cases:

    * If the tumor has not been treated for at least 5 years or is in a disease-
    * At least one year has elapsed since complete resection of basal cell cancer/flat cell cancer or successful treatment of cervical intraepithelial cancer
20. Patients with genetic problems such as galactose intolerance, Laplactase deficiency or glucose-galactose malabsorption
21. Patients with acute diffuse invasive lung disease and heart disease
22. Patients with history of hypersensitivity to Lenalidomide and bortezomib

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
3-Year Progression-free survival (PFS) | 3-years after randomization
  The time from randomization into the date of first observation of documented disease progression or death.

SECONDARY OUTCOMES:
Assessment of response | accessed every each cycle (each cycle is 28days)
  Response will be determined by the International Myeloma Working Group Response Criteria every cycle

OTHER OUTCOMES:
Minimal residual disease (MRD) | at the time when patient get CR or VGPR after 1year administration
  Confirmation of MRD negativity

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided